CLINICAL TRIAL: NCT04563897
Title: Contrast-enhanced Ultrasound in Liver Tumor by Sonazoid
Brief Title: Prospective Multicenter Study on Clinical Application of Sonazoid in Liver Tumor
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Ping Liang, Department of Interventional Ultrasound, Chinese PLA General Hospital
Other Study IDs: S2020-300-03
Record Dates: First submitted 2020-09-21; First posted 2020-09-25 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Ultrasound
Keywords: Focal liver lesions

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- HBV/HCV
- Fatty liver disease
- Liver background after systematic treatment
- normal hepatic background

SUMMARY:
Sonazoid as a new generation of ultrasound contrast agent.This study based on the features of Sonazoid specific angiography and his mechanical index, the role of Sonazoidin in the differential diagnosis of benign and malignant focal liver lesions in different liver background was explored

DETAILED DESCRIPTION:
Sonazoid as a new generation of ultrasound contrast agent, was liver specificity (Kupffer cells), macrophages at the very stable period, Kupffer imaging contrast enhancement effect for more than 1 hour, it is mainly used for focal liver lesions of blood vessels and Kupffer phase of ultrasonic imaging, facilitate early detection of small lesions (< 1 cm). Until now, Sonazoid has been mainly focused on liver focal lesions.

Most liver cancer patients in China are associated with chronic liver disease, and more than 80% of liver disease patients are in advanced stage at the time of treatment. Differential diagnosis is still a challenge for enhanced CT / MRI. About 40% of HCCs lack arterial phase enhancement and 40% - 60% of small lesions do not show elution in venous phase. The existing imaging methods have low sensitivity in detecting small lesions, and it is difficult to detect lesions smaller than 1 cm. Studies have found that the sensitivity of CT and MRI is of 60 - 94.4% and 58.5 - 93% respectively when the tumor diameter is larger than 1 cm. When the tumor diameter is less than 1 cm, the sensitivity of CT and MRI to detect tumors is reduced to 33 - 45% and 33 - 67%, respectively. The diagnostic efficiency of conventional ultrasonography for small lesions, especially in patients with chronic hepatitis B or cirrhosis, is poor. Although the diagnostic efficiency of conventional contrast-enhanced ultrasound in the diagnosis of small lesions with chronic hepatitis B or liver cirrhosis has a certain improvement, there is still a large rate of missed diagnosis. In addition, ordinary ultrasound, conventional contrast-enhanced ultrasound, CT and MRI are very poor in the diagnosis of liver cancer differentiation, especially for highly differentiated liver cancer.

Sonazoid is a second generation ultrasound contrast agent, which is composed of microbubbles containing chemically stable and insoluble Perfluorobutane (PFB) gas and a hard shell of phosphatidylserine sodium (2-3 μ m in diameter) wrapped in the outer layer. These microbubbles can generate stable nonlinear oscillations in a low-power acoustic field and generate echoes at the second harmonic frequency of the transmitted pulse for enhanced contrast harmonic imaging . In addition to the ability of real-time angiography, Sonazoid microbubbles can be engulfed by Kupffer cells in the intrahepatic reticuloendothelial system to produce liver parenchymal imaging Usually 10 minutes after intravenous injection of Sonazoid contrast agent, Kupffer phase image appears, and normal liver parenchyma is enhanced . Therefore, at this stage, malignant lesions with little or no Kupffer cells are clearly demonstrated due to the lack of contrast media. In addition, because Sonazoid microbubbles can resonate without rupture under moderate ultrasonic pressure, Kupffer phase (Kupffer phase) imaging can be stable for more than several hours, which is beneficial to whole liver scanning . Because Sonazoid has the advantages of ultra long time development and good stability, Sonazoid has significant clinical advantages in the diagnosis of small liver cancer lesions, liver cirrhosis background liver cancer and highly differentiated liver cancer.. However, these studies based on Sonazoid are all small sample studies and subjective qualitative differential diagnosis methods, and lack of systematic analysis and research. Therefore, based on the advantages of the new ultrasound contrast agent, using qualitative analysis and quantitative analysis method to collect large samples, systematically explore the standardized diagnosis scheme and diagnostic efficiency of liver cancer with different liver background, which has important clinical significance for early diagnosis, early detection and improving the accuracy of diagnosis of liver cancer.

ELIGIBILITY:
Inclusion Criteria:

* 1.Chinese citizen, ≥ 18 years old; 2.Conventional ultrasound shows that there is definite lesion in the liver, and there is liver parenchyma around the lesion; 3.There is enhanced MRI or enhanced CT finding. For patients with liver fibrosis after hepatitis, the results of liver parenchyma elastography can be added (optional); 4. If the subjects are female, they should be non pregnant and lactating women; 5.Patients voluntarily participate in the study and signe informed consent

Exclusion Criteria:

* 1.Subjects are known to be allergic to Perfluorobutane or any component of Sonazoid; 2.Patients with severe heart disease or severe lung disease; 3.Pregnant, potential pregnant or lactating patients; 4.No enhanced MRI or CT results are available; 5.The researchers consider that the subjects are not suitable for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with definite liver neoplastic lesions, containing multiple kinds of liver background
Sampling Method: Non-Probability Sample
Enrollment: 1300 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2021-05-01 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance of contrast-enhanced ultrasound in different liver background and liver turmors by sonazoid | 10 months